CLINICAL TRIAL: NCT01654146
Title: An International Phase III Randomised Trial of Dose Fractionated Chemotherapy Compared to Standard Three Weekly Chemotherapy, Following Immediate Primary Surgery or as Part of Delayed Primary Surgery, for Women With Newly Diagnosed Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: ICON8: Weekly Chemotherapy in Ovarian Cancer
Acronym: ICON8
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Research Council (Other Government)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor-Investigator, Medical Research Council, Medical Research Council, Medical Research Council
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-022209-16; 10356387 (Other: ISRCTN)
Record Dates: First submitted 2012-06-20; First posted 2012-07-31 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; Epithelial ovarian carcinoma; Fallopian tube carcinoma; Primary serous peritoneal carcinoma; Gynaecological carcinoma; Randomised controlled trial
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Control Arm) (Active Comparator): Carboplatin and paclitaxel on day 1 of a 21-day cycle for 6 cycles
  Interventions: Drug: Carboplatin; Drug: Paclitaxel
- Arm 2 (Research arm) (Experimental): Carboplatin on day 1 and dose-fractionated weekly paclitaxel on day 1, 8 and 15 of a 21-day cycle for 6 cycles
  Interventions: Drug: Carboplatin; Drug: Paclitaxel
- Arm 3 (Research arm) (Experimental): Dose-fractionated weekly carboplatin and weekly paclitaxel on day 1, 8 and 15 of a 21-day cycle for 6 cycles.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Carboplatin — AUC5 by intravenous infusion over 30-60 minutes
  Arms: Arm 1 (Control Arm); Arm 2 (Research arm)
Drug: Carboplatin — AUC2 by intravenous infusion over 30-60 minutes
  Arms: Arm 3 (Research arm)
Drug: Paclitaxel — 175mg/m2 by intravenous infusion over 3 hours
  Arms: Arm 1 (Control Arm)
Drug: Paclitaxel — 80mg/m2 by intravenous infusion over 1 hour
  Arms: Arm 2 (Research arm); Arm 3 (Research arm)

SUMMARY:
The purpose of this study is to determine if weekly chemotherapy (i.e. giving paclitaxel or carboplatin at a lower dose every week) is more effective than standard chemotherapy (paclitaxel and carboplatin given once every three weeks over 18 weeks) in treating ovarian cancer. The investigators also want to see if weekly chemotherapy causes more or fewer side-effects than standard chemotherapy.

DETAILED DESCRIPTION:
ICON8 is a three-arm, three stage trial. Patients will be randomised in a 1:1:1 ratio. Patients in arm 1 (control arm) will receive weekly carboplatin and paclitaxel on day 1 of a 21-day cycle for 6 cycles. Patients in arm 2 will receive carboplatin on day 1 and dose-fractionated weekly paclitaxel on day 1, 8 and 15 of a 21-day cycle for 6 cycles. Patients in arm 3 will receive dose-fractionated weekly carboplatin and dose-fractionated weekly paclitaxel on day 1, 8 and 15 of a 21-day cycle for 6 cycles.

The trial will have three planned stages. Stage 1 will be conducted to confirm feasibility and safety of protocol treatment in all patients and separately in the Delayed Primary Surgery (DPS) patients. The outcome measure for stage 2 will be 9-month progression-free survival (PFS) rate. The primary outcome measures for stage 3 will be PFS and overall survival and secondary outcomes will be toxicity, Quality of Life and Health Economics. If pre-defined levels of deliverability, at stage 1, or activity, at stage 2, are not met then the research arms will be reconsidered.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 years or more
* Signed informed consent and ability to comply with the protocol
* Histologically confirmed, with core biopsy from a disease site as minimum requirement (cytology alone is insufficient for diagnosis):

  * Epithelial ovarian carcinoma
  * Primary peritoneal carcinoma of Müllerian histological type
  * Fallopian tube carcinoma
* FIGO stage IC or above, which may be based on clinical and radiological assessment in patients who have not undergone immediate primary surgery
* Confirmed high-risk histological subtype for patients with FIGO stage IC/IIA disease, namely:

  * High grade serous carcinoma
  * Clear cell carcinoma
  * Other histological subtype considered poorly differentiated/grade 3
* ECOG Performance Status (PS) 0-2
* Life expectancy > 12 weeks
* Adequate bone marrow function:

  * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/l
  * Platelets (Plt) ≥ 100 x 109/l
  * Haemoglobin (Hb) ≥ 9g/dl (can be post transfusion)
* Adequate liver function (within 28 days prior to randomisation):

  * Serum bilirubin (BR) ≤ 1.5 x ULN
  * Serum transaminases ≤ 3 x ULN in the absence of parenchymal liver metastases or ≤ 5 x ULN in the presence of parenchymal liver metastases
* Adequate renal function as defined by GFR (Glomerular Filtration Rate) ≥ 30ml/min.

Exclusion Criteria:

* Non-epithelial ovarian cancer, including malignant mixed Müllerian tumours (carcinosarcomas)
* Peritoneal cancer that is not of Müllerian origin, including mucinous histology
* Borderline tumours (tumours of low malignant potential)
* Prior systemic anti-cancer therapy for ovarian cancer (for example chemotherapy, monoclonal antibody therapy, tyrosine kinase inhibitor therapy or hormonal therapy)
* Previous malignancies within 5 years prior to randomisation apart from: adequately treated carcinoma in-situ of the cervix, breast ductal carcinoma in-situ, non-melanomatous skin cancer; or previous/synchronous early-stage endometrial cancer defined as stage IA (FIGO 2009) grade 1 or 2 endometrioid cancers with no lymphovascular space invasion
* Pre-existing sensory or motor neuropathy grade ≥ 2
* Evidence of any other disease/metabolic dysfunction that in the opinion of the investigator would put the subject at high-risk of treatment-related complications or prevent compliance with the trial protocol
* Planned intraperitoneal cytotoxic chemotherapy
* Any previous radiotherapy to the abdomen or pelvis
* Sexually active women of childbearing potential not willing to use adequate contraception (e.g. oral contraceptives, intrauterine device or barrier method of contraception in conjunction with spermicidal jelly or surgically sterile) for the study duration and at least six months afterwards
* Pregnant or lactating women
* Treatment with any other investigational agent prior to protocol defined progression
* Known hypersensitivity to carboplatin, paclitaxel or their excipients (including cremophor)
* History or clinical suspicion of brain metastases or spinal cord compression. CT/MRI of the brain is mandatory in the case of suspected brain metastases. Spinal MRI is mandatory in the case of suspected spinal cord compression. Patients with brain or meningeal metastases are not eligible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1485 (Estimated)
Dates: Start 2011-06; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Feasibility assessed as the number of cycles and dose intensity of protocol treatment delivered per patient. | 6 months after the 50th patient has been randomised to each arm and 6 months after the 50th patient with a plan to undergo delayed primary surgery has been randomised to each arm
Stage 1: Safety assessed as the rate of any ≥ grade 3 toxicity experienced per patient. | 6 months after the 50th patient has been randomised to each arm and 6 months after the 50th patient with a plan to undergo delayed primary surgery has been randomised to each arm
Stage 2: Progression Free Survival rate at 9 months after randomisation | 9 months after first 62 patients randomised per arm
Stage 3: Progression Free Survival | PFS expected 1 year after last patient is randomised. OS expected 3 years after last patient is randomised.
Stage 3: Overall Survival | PFS expected 1 year after last patient is randomised. OS expected 3 years after last patient is randomised.

SECONDARY OUTCOMES:
Stage 3: Toxicity assessed by number of participants with adverse events | Expected 1 year and 3 years after last patient is randomised.
  Assessment of toxicity profile of dose-fractionated chemotherapy
Stage 3: Quality of Life | Expected 1 year and 3 years after last patient is randomised.
  Assessment of potential impact of dose-fractionated chemotherapy on functionality and well-being in patients undergoing first line treatment for ovarian cancer.
Stage 3: Health Economics | Expected 1 year and 3 years after last patient is randomised.
  Cost-effectiveness analysis of dose-fractionated chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Research Council Clinical Trials Unit, London, United Kingdom

REFERENCES:
- [Derived] Colomban O, Clamp A, Cook A, McNeish IA, You B. Benefit From Fractionated Dose-Dense Chemotherapy in Patients With Poor Prognostic Ovarian Cancer: ICON-8 Trial. JCO Clin Cancer Inform. 2023 Apr;7:e2200188. doi: 10.1200/CCI.22.00188. PMID 37075255
- [Derived] Clamp AR, James EC, McNeish IA, Dean A, Kim JW, O'Donnell DM, Gallardo-Rincon D, Blagden S, Brenton J, Perren TJ, Sundar S, Lord R, Dark G, Hall M, Banerjee S, Glasspool RM, Hanna CL, Williams S, Scatchard KM, Nam H, Essapen S, Parkinson C, McAvan L, Swart AM, Popoola B, Schiavone F, Badrock J, Fananapazir F, Cook AD, Parmar M, Kaplan R, Ledermann JA. Weekly dose-dense chemotherapy in first-line epithelial ovarian, fallopian tube, or primary peritoneal cancer treatment (ICON8): overall survival results from an open-label, randomised, controlled, phase 3 trial. Lancet Oncol. 2022 Jul;23(7):919-930. doi: 10.1016/S1470-2045(22)00283-2. Epub 2022 Jun 9. PMID 35690073
- [Derived] Morgan RD, McNeish IA, Cook AD, James EC, Lord R, Dark G, Glasspool RM, Krell J, Parkinson C, Poole CJ, Hall M, Gallardo-Rincon D, Lockley M, Essapen S, Summers J, Anand A, Zachariah A, Williams S, Jones R, Scatchard K, Walther A, Kim JW, Sundar S, Jayson GC, Ledermann JA, Clamp AR. Objective responses to first-line neoadjuvant carboplatin-paclitaxel regimens for ovarian, fallopian tube, or primary peritoneal carcinoma (ICON8): post-hoc exploratory analysis of a randomised, phase 3 trial. Lancet Oncol. 2021 Feb;22(2):277-288. doi: 10.1016/S1470-2045(20)30591-X. Epub 2020 Dec 22. PMID 33357510
- [Derived] Blagden SP, Cook AD, Poole C, Howells L, McNeish IA, Dean A, Kim JW, O'Donnell DM, Hook J, James EC, White IR, Perren T, Lord R, Dark G, Earl HM, Hall M, Kaplan R, Ledermann JA, Clamp AR. Weekly platinum-based chemotherapy versus 3-weekly platinum-based chemotherapy for newly diagnosed ovarian cancer (ICON8): quality-of-life results of a phase 3, randomised, controlled trial. Lancet Oncol. 2020 Jul;21(7):969-977. doi: 10.1016/S1470-2045(20)30218-7. PMID 32615110